CLINICAL TRIAL: NCT00971308
Title: Open Label, Multiple-Dose Study to Evaluate the Antiviral Activity, Safety, Tolerability and Pharmacokinetics of BMS-824393 in Treatment Naive Subjects Infected With Hepatitis C Virus Genotype 1
Brief Title: Multiple Dose Study In Treatment Naive Subjects Infected With Hepatitis C Virus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI451-002
Record Dates: First submitted 2009-09-02; First posted 2009-09-03 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2011-01

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- BMS-824393 (Panel 1) (Experimental)
  Interventions: Drug: BMS-824393
- BMS-824393 (Panel 2) (Experimental)
  Interventions: Drug: BMS-824393
- BMS-824393 (Panel 3) (Experimental)
  Interventions: Drug: BMS-824393
- BMS-824393 (Panel 4) (Experimental)
  Interventions: Drug: BMS-824393
- BMS-824393 (Panel 5) (Experimental)
  Interventions: Drug: BMS-824393

INTERVENTIONS:
Drug: BMS-824393 — Capsule, Oral, 50mg, Once Daily, 3 days
  Arms: BMS-824393 (Panel 1)
Drug: BMS-824393 — Capsule, Oral, 100mg, Once Daily, 3 days
  Arms: BMS-824393 (Panel 2)
Drug: BMS-824393 — Capsule, Oral, 10mg, Once Daily, 3 days
  Arms: BMS-824393 (Panel 3)
Drug: BMS-824393 — Capsule. Oral, 1mg, Once Daily, 3 days
  Arms: BMS-824393 (Panel 4)
Drug: BMS-824393 — Capsule, Oral, Flexible, ≤100mg, Once Daily, 3 days
  Arms: BMS-824393 (Panel 5)

SUMMARY:
The purpose of this study is to determine the antiviral effect following three days of dosing with BMS-824393 in chronically genotype subtype 1a and 1b Hepatitis C virus (HCV) infected subjects.

ELIGIBILITY:
Inclusion Criteria:

* Treatment naive chronically infected subjects with Hepatitis C Virus genotype 1
* HCV RNA viral load of ≤10*5* IU/mL (100,000 IU/mL)
* Body Mass Index (BMI) of 18 to 35 kg/m², inclusive

Exclusion Criteria:

* Women who are pregnant or breast feeding
* Any significant acute or chronic medical illness which is not stable or is not controlled with medication or is not consistent with Hepatitis C infection
* Any other medical, psychiatric and/or social reason which, in the opinion of the Investigator, would make the candidate inappropriate for participation in this study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2009-10; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HCV RNA following three days of dosing with BMS-824393 in chronically genotype subtype 1a and 1b HCV infected subjects | On Days 1, 2, 3, 4, 5, 6, 7, 14, 28, 90 and 180 days after study drug administration

SECONDARY OUTCOMES:
To assess the change in HCV RNA over time during three days of dosing with BMS- 824393 and during the follow-up period in chronically genotype subtype 1a and 1b HCV infected subjects | On Days 1, 2, 3, 4, 5, 6, 7, 14, 28, 90 and 180 days after study drug administration
To assess potential differences in antiviral effect in genotype subtypes (1a versus 1b) | On Days 1, 2, 3, 4, 5, 6, 7, 14, 28, 90 and 180 days after study drug administration
To assess the safety and tolerability of multiple oral doses of BMS-824393 | On Days 1, 2, 3, 4, 5, 6, 7, 14, 28, 90 and 180 days after study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (6):
- United States (6):
  - Advanced Clinical Research Institute, Anaheim, California
  - West Coast Clinical Trials, Llc, Cypress, California
  - Elite Research Institute, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Parexel International - Baltimore Epcu, Baltimore, Maryland
  - Alamo Medical Research, San Antonio, Texas

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx